CLINICAL TRIAL: NCT02082808
Title: A Phase 1, Open-Label, Crossover Study to Evaluate the Drug Interaction Between Dolutegravir and Daclatasvir in Healthy Adult Subjects
Brief Title: Study to Evaluate the Drug Interaction Between Dolutegravir (DTG) and Daclatasvir (DCV) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201102
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Dolutegravir; healthy volunteer; pharmacokinetics; daclatasvir; drug interaction
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Participants will receive the study Treatment A for 5 days (DTG 50mg q24h) in Period 1 followed by a washout period (>=7days) and Treatment B for 5 days (DCV 60mg q24h) in Period 2 and Treatment C (DCV 60mg q24h + DTG 50mg q24h) for 5 days in Period 3
  Interventions: Drug: DTG; Drug: DCV
- Sequence 2 (Experimental): Participants will receive the study Treatment B for 5 days (DCV 60mg q24h) in Period 1 followed by a washout period (>=7days) and Treatment A for 5 days (DTG 50mg q24h) in Period 2 and Treatment C (DCV 60mg q24h + DTG 50mg q24h) for 5 days in Period 3
  Interventions: Drug: DTG; Drug: DCV

INTERVENTIONS:
Drug: DTG — DTG is provided as 9 millimetre white, film-coated, round tablets debossed with SV 572 on one side and 50 on the other side
Drug: DCV — DCV is provided as a plain, green, biconvex, pentagonal film-coated tablet

SUMMARY:
This study is designed to estimate the two-way drug interaction between DCV and DTG as a drug interaction between DTG and DCV is expected to be low and this study is to be performed as confirmation. This will be a single-center, open-label, three-period, crossover study in healthy adult subjects. This study to describe and compare steady-state plasma DTG and DCV pharmacokinetics following administration of DTG 50 mg q24h with and without DCV 60 mg q24h and following administration of DCV 60 mg q24h with and without DTG 50 mg q24h also the safety and tolerability was assessed after a repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and after a repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with serum creatinine values outside the normal range should always be excluded from enrollment.
* Body weight >=50 kg for males and 45 kg for females and BMI within the range 18.5-31.0 kg/m^2 (inclusive).
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit/mL and estradiol <40 picogram/mL (<147 picomolar/L) is confirmatory.

Child-bearing potential with negative pregnancy test as determined by serum or urine hCG test at screening or prior to dosing AND Agrees to use the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 72 hours post the last dose.

OR has only same-sex partners, when this is her preferred and usual lifestyle.

* Male subjects with female partners of child-bearing potential must agree to use the contraception methods. This criterion must be followed from the time of the first dose of study medication until 72 hours post the last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase, alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTc <450 msec

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus antibody.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters of DTG following DTG 50 mg q24h administration with and without DCV 60mg q24h | Day 5 in Period 1 or 2, and Period 3: pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 8, 12 and 24 hours post morning dose
  Plasma PK parameters for DTG include steady state area under the concentration-time curve over the dosing interval (AUC (0-tau)), maximum observed concentration (Cmax), concentration at the end of the dosing interval (Ctau), apparent clearance following oral dosing (CL/F) and terminal phase half-life (t1/2) , following DTG 50 mg q24h administration with and without DCV 60mg q24h
Composite of PK parameters of DCV following administration of DCV 60 mg q24h with and without DTG 50 mg q24h | Day 5 (Periods 1 or 2, and Period 3): pre-dose (within 15 minutes prior to dosing), 0.5,1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24hrs post morning dose
  Plasma DCV steady state AUC(0-tau), Cmax, Ctau, CL/F and t1/2 following administration of DCV 60 mg q24h with and without DTG 50 mg q24h

SECONDARY OUTCOMES:
Safety and Tolerability of DTG and DCV as assessed by adverse event | Up to 36 days
  Safety and tolerability of repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h will be assessed by adverse events
Safety and Tolerability of DTG and DCV as assessed by concurrent medication | Up to 36 days
  Safety and tolerability of repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h will be assessed by concurrent medication
Safety and Tolerability of DTG and DCV as assessed by clinical laboratory | Up to 36 days
  Safety and tolerability of repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h will be assessed by clinical laboratory
Safety and Tolerability of DTG and DCV as assessed by ECG | Screening
  Safety and tolerability of repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h will be assessed by ECG
Safety and Tolerability of DTG and DCV as assessed by vital signs assessments | Up to 36 days
  Safety and tolerability of repeat dose DTG 50 mg q24h with or without DCV 60 mg q24h and repeat dose DCV 60 mg q24h with and without DTG 50 mg q24h will be assessed by vital signs assessments (blood pressure and heart rate)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Ross LL, Song IH, Arya N, Choukour M, Zong J, Huang SP, Eley T, Wynne B, Buchanan AM. No clinically significant pharmacokinetic interactions between dolutegravir and daclatasvir in healthy adult subjects. BMC Infect Dis. 2016 Jul 22;16:347. doi: 10.1186/s12879-016-1629-5. PMID 27450277